CLINICAL TRIAL: NCT07055867
Title: Epidemiological and Clinical Characteristics of Mpox Outbreak in Equateur, the DR Congo (Part1)
Status: Enrolling by invitation | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Principal Investigator, Yasutoshi KIDO, Professor, Osaka Metropolitan University
Other Study IDs: N553/BN/PMMF/2024
Record Dates: First submitted 2025-05-06; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mpox (Monkeypox)
Keywords: test negative control; case control; outbreak investigation; Mpox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Skin lesion and oral mucosa swab sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Cases are defined as Individuals who reported to local health agents with symptoms consistent with mpox and subsequently tested positive for mpox through a molecular-based diagnostic test.
- Control: Controls are defined as Individuals who reported to local health agents with symptoms consistent with mpox but subsequently tested negative for mpox through a molecular-based diagnostic test. Among individuals with a negative molecular diagnostic test for mpox, those who have passed more than 21 days since the onset of mpox-like signs and symptoms or those whom serological testing confirms prior exposure to mpox will be excluded as controls from analysis to avoid confounding results.
  Rationale: It is not possible to reliably distinguish between uninfected individuals and convalescents. Previous studies suggest a median recovery time of approximately 21 days.

SUMMARY:
The goal of this observational study is to characterize the clinical features of the 2024 mpox outbreak in Equateur Province of DRC and to identify associated risk factors. The main question it aims to answer is:

* What are the clinical features of the 2024 mpox outbreak in Equateur Province of DRC?
* What are the associated risk factors of the 2024 mpox outbreak? Participants which has mpox like symptoms will answer mpox investigations related questions and be collected skin lesions and whole blood samples.

DETAILED DESCRIPTION:
Mpox is caused by the monkeypox virus (MPXV), a member of the genus Orthopoxvirus (family Poxviridae). This virus is closely related to the variola virus, which causes smallpox. MPXV was first identified in 1958, and the first human case was reported in the Democratic Republic of the Congo (DRC) in 1970. It was presumed that the smallpox (vaccinia) vaccine would confer cross-protection against mpox. Following the global eradication of smallpox in 1980, mpox remained largely confined to limited regions in Central Africa-where zoonotic spillover from wild animal reservoirs constituted the primary route of transmission. Equateur Province is among the areas in the DRC with a notably high burden of reported mpox cases.

Over the past five decades, routine smallpox vaccination ceased worldwide, resulting in waning herd immunity against orthopoxviruses. During this period, mpox incidence rose markedly, with an estimated tenfold increase in global cases. Two principal genetic clades of MPXV have been identified: clade I (historically referred to as the Congo Basin clade) and clade II (the West African clade). In 2018, Nigeria experienced a resurgence of mpox, highlighting the virus's potential to emerge in previously controlled areas. Starting in 2022, clade II mpox circulated globally, especially among men who have sex with men (MSM), peaking in mid-2022 before declining to persistently lower levels by early 2023. Although clade II mpox typically exhibits a low case-fatality ratio (<1%), clade I has historically been associated with more severe disease and higher mortality. In 2023, the number of reported mpox cases continued to climb in the DRC, prompting the World Health Organization (WHO) to declare a Public Health Emergency of International Concern (PHEIC) in August 2024.

Recent surveillance indicates that sub-clade Ia MPXV is spreading in western DRC through multiple transmission modes, including contact with infected wild animals, household exposure, or sexual contact. By contrast, sub-clade Ib mpox in the eastern part of the country appears initially to spread via intimate or sexual contact between adults, followed by household transmission. Numerous environmental and social risk factors-including the consumption of rodent species, deforestation, climate change, civil unrest, population displacement, emerging MPXV variants, and weakened immunity-may be driving mpox incidence. Clade Ia mpox is currently affecting western parts of the DRC, yet the epidemiology remains poorly understood due to the limited number of laboratory-confirmed cases.

This study aims to characterize the clinical features of the 2024 mpox outbreak in Equateur Province of DRC and to identify associated risk factors. The findings will advance understanding of mpox transmission dynamics and disease severity, ultimately informing more effective prevention and control strategies in endemic settings.

ELIGIBILITY:
Inclusion Criteria:

• Provision of informed consent: Proxy-assisted informed consent is allowed under safety considerations. Following oral consent, the investigator will document this on the informed consent form as a witness.

• Fulfillment of the current mpox clinical case definition in the DRC, which includes: Presence of a vesicular or pustular eruption with deep-seated, firm pustules.

At least one of the following symptoms:

Fever preceding the eruption. Lymphadenopathy (inguinal, axillary, or cervical). Presence of pustules or crusts on the palms of the hands or soles of the feet. • Laboratory confirmation: At least one molecular-based mpox diagnostic test confirming the diagnosis.

Exclusion Criteria:

Participants will be excluded from the study under the following conditions:

• Refusal to participate in the study: Individuals who decline to provide consent for study participation will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study targets patients reported as suspected mpox cases (all ages, both sexes) to the Health District Central Office in the selected sites. For participants aged under 15 years or those with impaired communication abilities (e.g., due to altered consciousness or severe medical conditions), consent must be obtained from a parent, legal guardian, or responsible caregiver. The study population is designed to minimize selection bias related to health-seeking behavior.
  All patients suspected of having mpox and who provide proxy-assisted written informed consent to participate in the study are eligible for inclusion due to reduction of the risk of contact transmission with verbal agreement documented and confirmed by a witness. This approach prioritizes participant and staff safety while adhering to ethical standards.
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mpox positivity | Day 1
  Mpox positivity is determined based on one or more molecular-based diagnostic tests. In addition to standard diagnostic methods, the study will assess the performance of novel diagnostic platforms, such as loop-mediated isothermal amplification (LAMP) assays. These platforms will be evaluated for sensitivity, specificity, and overall diagnostic accuracy compared to established molecular-based techniques.
Virological Course | Day1 and 3-4 weeks after baseline
  Genotypes and longitudinal changes in viral load (measured as copies/mL) will be monitored over multiple time points during the study period.
  Genotypes and quantitative viral load dynamics will reflect disease progression and the timeline of viral clearance, providing insights into the natural course of infection.
Disease outcome | Day1 and 3-4 weeks after baseline
  Mpox severity will be evaluated based on skin lesion burden, clinical complications, organ dysfunction, and mortality outcomes.
  Scoring Criteria:
  Mild: Fewer than 25 lesions. Moderate: 26-99 lesions. Severe: 100 or more lesions or the presence of organ dysfunction, regardless of lesion count.
  Fatal Outcome: If a patient dies from mpox or its complications during the study, the case will be classified as "fatal outcome." Assessment: The severity score will integrate the number of skin lesions across various anatomical sites and documented signs of complications (e.g., respiratory distress, neurological symptoms, renal impairment).
Serological Response | Day1 and 3-4 weeks after baseline
  The serological response will be assessed through the detection and quantification of mpox-specific antibodies(Arbitrary Unit) at different time points.
  Evaluate the kinetics of the humoral immune response during and after infection.
  Determine correlations between serological responses, disease severity, and virological clearance.

SECONDARY OUTCOMES:
Performance of Novel Diagnostic Platforms | Day 1
  To compare the performance of LAMP-based diagnostics and other emerging diagnostic methods with conventional molecular techniques like PCR.
  Outcome Metrics: Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and turnaround time.
Clinical Recovery | 3-4 weeks after baseline
  Defined by the resolution of symptoms and the absence of detectable viral load during follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Yasutoshi Kido, Professor, Principal Investigator — Osaka Metropolitan Unievrsity
Locations (1):
- Equateur Provincial Public Health Laboratory, Mbandaka, Équateur Province, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Z, Sinha A, Zhang Y, Tanner N, Cheng HT, Premsrirut P, Carlow CKS. Extraction-free LAMP assays for generic detection of Old World Orthopoxviruses and specific detection of Mpox virus. Sci Rep. 2023 Nov 30;13(1):21093. doi: 10.1038/s41598-023-48391-z. PMID 38036581
- [Background] Mazzotta V, Nozza S, Lanini S, Moschese D, Tavelli A, Rossotti R, Fusco FM, Biasioli L, Matusali G, Raccagni AR, Mileto D, Maci C, Lapadula G, Di Biagio A, Pipito L, Tamburrini E, Monforte AD, Castagna A, Antinori A; mpox-Icona study group. Clinical and laboratory predictors of mpox severity and duration: an Italian multicentre cohort study (mpox-Icona). EBioMedicine. 2024 Sep;107:105289. doi: 10.1016/j.ebiom.2024.105289. Epub 2024 Aug 22. PMID 39178746
- [Background] Osadebe L, Hughes CM, Shongo Lushima R, Kabamba J, Nguete B, Malekani J, Pukuta E, Karhemere S, Muyembe Tamfum JJ, Wemakoy Okitolonda E, Reynolds MG, McCollum AM. Enhancing case definitions for surveillance of human monkeypox in the Democratic Republic of Congo. PLoS Negl Trop Dis. 2017 Sep 11;11(9):e0005857. doi: 10.1371/journal.pntd.0005857. eCollection 2017 Sep. PMID 28892474
- [Background] Ozasa K, Fukushima W. Commentary: Test-Negative Design Reduces Confounding by Healthcare-Seeking Attitude in Case-Control Studies. J Epidemiol. 2019 Aug 5;29(8):279-281. doi: 10.2188/jea.JE20180177. Epub 2018 Nov 10. No abstract available. PMID 30416164
- [Background] Moraes-Cardoso I, Benet S, Carabelli J, Perez-Zsolt D, Mendoza A, Rivero A, Alemany A, Descalzo V, Alarcon-Soto Y, Grifoni A, Sette A, Molto J, Marc A, Marks M, Mitja O, Brander C, Paredes R, Izquierdo-Useros N, Carrillo J, Suner C, Olvera A, Mothe B; MoViE-Immune study group. Immune responses associated with mpox viral clearance in men with and without HIV in Spain: a multisite, observational, prospective cohort study. Lancet Microbe. 2024 Aug;5(8):100859. doi: 10.1016/S2666-5247(24)00074-0. Epub 2024 Jun 7. PMID 38857615
- [Background] CLINICAL MANAGEMENT AND INFECTION PREVENTION AND CONTROL FOR MONKEYPOX. 2022 https://iris.who.int/bitstream/handle/10665/355798/WHO-MPX-Clinical_and_IPC-2022.1-eng.pdf?sequence=1 (accessed Dec 7, 2024).
- [Background] Vakaniaki EH, Kacita C, Kinganda-Lusamaki E, O'Toole A, Wawina-Bokalanga T, Mukadi-Bamuleka D, Amuri-Aziza A, Malyamungu-Bubala N, Mweshi-Kumbana F, Mutimbwa-Mambo L, Belesi-Siangoli F, Mujula Y, Parker E, Muswamba-Kayembe PC, Nundu SS, Lushima RS, Makangara-Cigolo JC, Mulopo-Mukanya N, Pukuta-Simbu E, Akil-Bandali P, Kavunga H, Abdramane O, Brosius I, Bangwen E, Vercauteren K, Sam-Agudu NA, Mills EJ, Tshiani-Mbaya O, Hoff NA, Rimoin AW, Hensley LE, Kindrachuk J, Baxter C, de Oliveira T, Ayouba A, Peeters M, Delaporte E, Ahuka-Mundeke S, Mohr EL, Sullivan NJ, Muyembe-Tamfum JJ, Nachega JB, Rambaut A, Liesenborghs L, Mbala-Kingebeni P. Sustained human outbreak of a new MPXV clade I lineage in eastern Democratic Republic of the Congo. Nat Med. 2024 Oct;30(10):2791-2795. doi: 10.1038/s41591-024-03130-3. Epub 2024 Jun 13. PMID 38871006
- [Background] WHO Director-General declares mpox outbreak a public health emergency of international concern. Saudi Med J. 2024 Aug;45(9):1002-1003. No abstract available. PMID 39218470
- [Background] Besombes C, Mbrenga F, Malaka C, Gonofio E, Schaeffer L, Konamna X, Selekon B, Namsenei-Dankpea J, Gildas Lemon C, Landier J, von Platen C, Gessain A, Manuguerra JC, Fontanet A, Nakoune E. Investigation of a mpox outbreak in Central African Republic, 2021-2022. One Health. 2023 Jun;16:100523. doi: 10.1016/j.onehlt.2023.100523. Epub 2023 Mar 7. PMID 36950196
- [Background] Ladnyj ID, Ziegler P, Kima E. A human infection caused by monkeypox virus in Basankusu Territory, Democratic Republic of the Congo. Bull World Health Organ. 1972;46(5):593-7. PMID 4340218
- [Background] Thornhill JP, Barkati S, Walmsley S, Rockstroh J, Antinori A, Harrison LB, Palich R, Nori A, Reeves I, Habibi MS, Apea V, Boesecke C, Vandekerckhove L, Yakubovsky M, Sendagorta E, Blanco JL, Florence E, Moschese D, Maltez FM, Goorhuis A, Pourcher V, Migaud P, Noe S, Pintado C, Maggi F, Hansen AE, Hoffmann C, Lezama JI, Mussini C, Cattelan A, Makofane K, Tan D, Nozza S, Nemeth J, Klein MB, Orkin CM; SHARE-net Clinical Group. Monkeypox Virus Infection in Humans across 16 Countries - April-June 2022. N Engl J Med. 2022 Aug 25;387(8):679-691. doi: 10.1056/NEJMoa2207323. Epub 2022 Jul 21. PMID 35866746